CLINICAL TRIAL: NCT05459662
Title: A Randomized Cross-over Double Arm Control Trial Evaluating the Impact of the Daily Consumption of Plant-based Diversified Meal Over a 2 Weeks Period on the Adult Gut Microbiome
Brief Title: Impact of Consuming a Plant-based Enriched Meal on the Adult Gut Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2106NRC2
Record Dates: First submitted 2022-05-24; First posted 2022-07-15 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oat based porridge (Placebo Comparator): Oat based porridge prepared with 64g of oat, 200ml of milk and 10 g of honey by the participant and consumed orally daily for 14 days as breakfast replacement
  Interventions: Dietary Supplement: oat based porridge
- Enriched plant-based meal (Active Comparator): Enriched plant-based meal pots (400 g) mixed with 25g of seeds and nuts consumed orally daily for 14 days as breakfast replacement
  Interventions: Dietary Supplement: plant based preparation

INTERVENTIONS:
Dietary Supplement: oat based porridge — Consume one preparation per day, orally
  Arms: Oat based porridge
Dietary Supplement: plant based preparation — Consume one preparation per day, orally
  Arms: Enriched plant-based meal

SUMMARY:
The aim of this study is to evaluate the impact of a diversified plant-based meal on the gut microbiome and its composition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years,
* Healthy participants, both male and female,
* BMI in the normal and overweight range 18.5 ≤ BMI ≤ 29.9 kg/m2,
* Able to understand and to sign a written informed consent prior to study enrolment.

Exclusion Criteria:

* Known chronic diseases or conditions for which the investigators/investigation team deem as not suitable for study participation,
* Known food allergy and intolerance e.g. lactose intolerance, nuts allergy,
* Habitually, have < 5 spontaneous bowel movements on average per week,
* Chronic or recurrent diarrhoea with spontaneous bowel movements > 2 per day
* Prior gastrointestinal surgery (apart from appendectomy or herniotomy),
* Received systemic antiviral/antibacterial/antifungal therapy during the 3 months prior to study enrolment,
* Medications or supplements that are known to alter gut function or microflora i.e. acid antisecretory drugs, pre-/probiotics, laxative during the 4 weeks prior to study enrolment,
* Anti-hyperlipidaemic, antihypertensive medications and/or anticoagulant agents,
* Currently participating in another interventional clinical trial or research project,
* Alcohol intake > 2 servings per day; specifically, a serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of beer. Or other chronic substance abuse,
* Changing diet patterns due to travelling and staying abroad for more than two weeks (Asia, Africa, or Latin America) during the two months prior to study enrolment,
* Food restrictions such as vegan, vegetarian, ketogenic, low carb, paleo, raw diets, caloric restrictive diets,
* Artificially sweetened beverage intake >1000 ml/ per day,
* Female participants will be excluded if they are pregnant, have given birth in the last 6 months, or are lactating,
* Subject having a hierarchical or family link with the research team members,
* Occurrence of fever episodes, infection, or vaccination during 14 days before the start of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Microbiota diversity & composition | Throughout 14 days of product intake
  Measured by Next Generation Sequencing (NGS)

SECONDARY OUTCOMES:
Change in quality of life using SF-36 questionnaire (Short Form 36 Health Survey) | Throughout 14 days of product intake
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients. Score ranging from 0 to 100 (higher scores indicate better health status).
Change in Short Chain Fatty Acids (SCFA) in the stool | Throughout 14 days of product intake
  Measured using Gas Chromatography (GC)
Gastrointestinal Symptom Rating Scale (GSRS) | Throughout 14 days of product intake
  Validated questionnaire exploring the presence and severity of GI symptoms over the previous 7 days. The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting reflux, abdominal pain, indigestion, diarrhea and constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms. The effect of the interventions on the GSRS will be assessed by a linear mixed model and will take into account information on this from all 7 days of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Innovation Lab, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No